CLINICAL TRIAL: NCT06632665
Title: Effects of Transcutaneous Vagus Nerve Stimulation With Virtual Reality on Upper Limb Functions in Post-stroke Patients
Brief Title: Effects Of Transcutaneous Vagus Nerve Stimulation With Virtual Reality In Post-Stroke Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0230
Record Dates: First submitted 2024-10-08; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Stroke
Keywords: Hand dexterity,Quality of life,Stroke,Transcutaneous vagus nerve stimulation,Upper limb motor function, Virtual reality.
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Transcutaneous vagus nerve stimulation+Virtual Reality+Routine physical therapy (Experimental): Patients will undergo a 60-minute session for two weeks, consisting of 30 minutes of vagus nerve stimulation, 15 minutes of virtual reality training, and 15 minutes of routine physiotherapy for 4 weeks
  Interventions: Other: transcutaneous vagus nerve stimulation+virtual reality+routine physical therapy
- Group B: Transcutaneous Vagus Nerve Stimulation +Routine physical therapy (Experimental): Patients will undergo a 60-minute session for two weeks, which includes 30 minutes of vagus nerve stimulation and 30 minutes of routine physiotherapy per session for 4 weeks.
  Interventions: Other: transcutaneous vagus nerve stimulation+routine physical therapy

INTERVENTIONS:
Other: transcutaneous vagus nerve stimulation+virtual reality+routine physical therapy — Transcutaneous vagus nerve stimulation Location The left auricular branch vagus nerve will be stimulated by the modified dot -like electrodes will be fitted to the cymba conchae.frequency:Stimulation perform for 30 minutes per day for 4 weeks .
  duration 600 pulses (intratrain pulse) frequency =20 Hz ; Pulse duration =0.3ms ,lasting 30 seconds each time ,stimulating once every 5 minutes
  Arms: Group A: Transcutaneous vagus nerve stimulation+Virtual Reality+Routine physical therapy
Other: transcutaneous vagus nerve stimulation+routine physical therapy — Transcutaneous vagus nerve stimulation Location The left auricular branch vagus nerve will be stimulated by the modified dot -like electrodes will be fitted to the cymba conchae.Stimulation perform for 30 minutes per day for 4 weeks .
  Routine physical therapy Stretching Areas :upper chest ,neck flexors ,shoulder flexor and adductors ,elbow and wrist flexors 10 minute per session,and stretches will held for 10s -30swith four repetition of each.30 minutes per day for 4 weeks Upper extremity Proprioception ,coordination,speed and agility increase such as followReach and grasp Handle turning simulated eating task Inserting object Opening bottle strenghtening exercise Muscles biceps brachii brachialis Coracobrachialis triceps brachii wrist extensors 10 minute per session for 4 weeks
  Arms: Group B: Transcutaneous Vagus Nerve Stimulation +Routine physical therapy

SUMMARY:
Stroke is a neurological condition also known as cerebrovascular accident occurs when blood supply to the brain is disrupted ,either by blockage or rupture of a blood vessels. Upper limb impairment after a stroke denotes diminished function in the arm, hand, wrist, and fingers due to neurological damage. Virtual Reality and Trascutaneous vagus nerve stimulation are innovative for post-stroke upper limb rehabilitation VR enhances motor learning and engagement with exercises and feedback, while VNS boosts neuroplasticity and reduces inflammation via vagus nerve stimulation. The aim of the study is to determine the effects of transcutaneous vagus nerve stimulation with virtual reality and routine physiotherapy on upper limb motor function, hand dexterity function and quailty of life .

This randomized clinical trial will be conducted at Al Ehsan Welfare,Lahore .The sample size calculated for this trial will be 50 .The patients will be randomly allocated using online randomization tool into 2 groups. Group A will receive Transcutaneous vagus nerve stimulation with Virtual Reality and Routine physical therapy.Patients will undergo a 60-minute session for four weeks, consisting of 30 minutes of vagus nerve stimulation, 15 minutes of virtual reality training, and 15 minutes of routine physiotherapy for 4 weeks, Group B will receive Transcutaneous Vagus Nerve Stimulation with Routine physical therapy Patients will undergo a 60-minute session for four weeks, which includes 30 minutes of vagus nerve stimulation and 30 minutes of routine physiotherapy per session for 4 weeks.

Purdue pegboard test will be used to assess dexterity function,Fugl - meyer assesment FMA - UE to assess Motor function of upper extremity, Stroke impact scale to measure Quality of life.The assessment will be conducted by assessor at baseline, 2 weeks, 4 weeks, and during a follow-up at 8 weeks after discontinuation of in-clinic therapy.The p value will be set at P= 0.05 to reported any significant difference.Kolmogorov-smirnov test will be used to check the normality of data . For the between group analysis Independent t test will be applied for parametric and Mann Whitney test will be applied for non parametric data. For within group comparison repeated measure ANOVA and Friedman ANOVA will be applied for parametric and non parametric data

ELIGIBILITY:
Inclusion Criteria:

* Patients with ischemic stroke at least more than 6 months.
* Patients having Montreal Cognitive Assessment (MoCA) score 26/30
* Patients able to follow and accept verbal instruction
* patients with normal sympathetic acitivity.

Exclusion criteria:

* Patients with history of previous surgical intervention on vagus nerve
* Patients having low heart rate 60 bpm
* Patients with history of any visual and hearing problem
* Patients with history of neuromuscular disorder affecting the function of upper limbs .
* Patients with advance liver,kidney,cardiac ,pulmonary disease
* Patients with history of orthopedic surgery and botulinum toxin injection.
* Patients with increase sympathetic activity.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-10-05 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment (FMA) | 4th week
  The Fugl-Meyer Assessment is a well established and effective clinical tool designed to assess motor function in individual extensively validated in stroke patients.
Purdue pegboard test | 4th week
  Purdue pegboard test The Purdue Pegboard Test developed by Joseph Tiffin in 1948 ,is widely utilized by clinicians and researchers to assess both gross movementand fingertip dexterity of the arm,hand,and fingers. It consist of a board with 4 cups across the top,containing pegs ,collars,and washers, and two vertical rows of 25 small holes down the center .This test is particularly suitable for evaluating patients with upper extremity impairments caused by neurological or musculoskeletal conditions.
Stroke Impact Scale | 4th week
  The Stroke Impact Scale is a comprehensive assessment tool designed by Duncan et al.specifically for measuring various aspects of health related quality of life in strokes survivors.it consists of 59 items ,each rated on a 5-point likert scale to gauge the level of difficulty experienced by patients.scores are aggregated into different domains ,with a standardized scoring system ranging from 0 to 100 .higher scores reflect a better quality of life across different dimensions impacted by stoke

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, PhD-PT, Study Chair — Riphah International University

IPD SHARING:
Plan to Share IPD: No